CLINICAL TRIAL: NCT03033342
Title: Randomized, Double-Blind, Placebo-Controlled Three-Part Phase 1 Study of Safety, Tolerability, Pharmacokinetics, and Food Effect of MRX-4 Administered Orally to Healthy Volunteers in Single and Multiple Ascending Dose Cohorts to Evaluate Drug Interactions With Omeprazole
Brief Title: Single Dose and Multiple Dose Escalation Trial of an Oral Formulation of MRX-4
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MicuRx (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: MRX4-001
Record Dates: First submitted 2016-12-19; First posted 2017-01-26 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2017-09

CONDITIONS: Safety
Keywords: Phase 1
MeSH Terms: interventions — Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Oral single doses of MRX-4 (Experimental): Single escalating oral doses of MRX-4 from 250 mg to 3000 mg
  Interventions: Drug: Oral single doses of MRX-4
- Oral multiple doses of MRX-4 (Experimental): Twice daily escalating oral doses of MRX-4 for 10 days: 500 mg, 750 mg, 1000 mg, and 1500 mg
  Interventions: Drug: Oral multiple doses of MRX-4
- MRX-4 co-administered with omeprazole (Experimental): Impact of concomitant food or omeprazole on the pharmacokinetics of oral MRX-4.
  Interventions: Drug: MRX-4 co-administered with omeprazole
- Oral single doses of placebo (Placebo Comparator): Single oral doses of placebo to match MRX-4
  Interventions: Drug: Oral single doses of placebo
- Oral multiple doses of placebo (Placebo Comparator): Multiple oral doses of placebo given twice daily for 10 days to match MRX-4
  Interventions: Drug: Oral multiple doses of placebo
- Placebo co-administered with omeprazole (Placebo Comparator): Oral placebo given on Day 1, Day 7 to match MRX-4 dosing with omeprazole
  Interventions: Drug: Placebo co-administered with omeprazole

INTERVENTIONS:
Drug: Oral single doses of MRX-4 — Oral single escalating doses of MRX-4
  Arms: Oral single doses of MRX-4
Drug: Oral multiple doses of MRX-4 — Multiple ascending doses of MRX-4 given twice daily for 10 days
  Arms: Oral multiple doses of MRX-4
Drug: MRX-4 co-administered with omeprazole — MRX-4 given orally on Day 1 and Day 7, co-administered with omeprazole on Day 3 through Day 7
  Arms: MRX-4 co-administered with omeprazole
Drug: Oral single doses of placebo — Single doses of placebo to match MRX-4
  Arms: Oral single doses of placebo
Drug: Oral multiple doses of placebo — Oral placebo given twice daily for 10 days to match the oral MRX-4
  Arms: Oral multiple doses of placebo
Drug: Placebo co-administered with omeprazole — Placebo given orally on Day 1 and Day 7, co-administered with omeprazole on Day 3 through Day 7
  Arms: Placebo co-administered with omeprazole

SUMMARY:
A phase one study of the safety, tolerability, and pharmacokinetics of a new oxazolidinone antibiotic. Cohorts of healthy adults (female and male) will participate in:

single dose escalation study of increasing doses of MRX-4 given by mouth others will participate in multiple dose escalation cohorts of MRX-4 given twice daily by mouth.

other cohorts of subjects will participate in the study to evaluate the impact of concomitant food or Omeprazole on safety, tolerability and pharmacokinetics of MRX-4

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Underlying hepatic, renal, metabolic, hematologic, cardiovascular, or immunologic disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2016-08-02 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-02-01 (Actual)

PRIMARY OUTCOMES:
Safety of single and multiple ascending doses of MRX-4 | Screening through end of study visit on Day 7 (Part 1), Day 17 (Part II) and Day 14 (Part III)
  Summary of number of subjects with changes in vital signs, physical examinations, clinical lab data, ECG parameters and adverse events
Summary of concentration time data for MRX-4 and its metabolites | Pre-dose through 72 hours post dose
  Concentration time data for MRX-4 and its metabolites in blood and urine

SECONDARY OUTCOMES:
Summary of the plasma concentration teim data for MRX-4 under fed or fasted conditions | Pre-dose through 72 hours post dose
  Concentration time data for MRX-4 and its metabolites in blood and urine under fed and fasted conditions
Safety of MRX-4 co-administered with omeprazole | Screening through end of study on Day 14
  Summary of the number of subjects with changes in vital signs, physical examinations, clinical lab data, ecg parameters and adverse events
Summary of the plasma concentration time data for MRX-4 co-administered with omeprazole | Pre-dose through 72 hours post dose
  Concentation time data for MRX-4 and its metabolites in blood and urine with and without omeprazole

IPD SHARING:
Plan to Share IPD: No
The study results will be published in the future